CLINICAL TRIAL: NCT06945237
Title: A Randomized Controlled Study on the Efficacy and Safety of Gut-Brain Neuromodulators in Patients With Gastroesophageal Reflux Disease
Brief Title: Efficacy of Gut-Brain Neuromodulators in the Treatment of Gastroesophageal Reflux Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, Shengliang Chen, Professor, RenJi Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RJYYQKLY-04
Record Dates: First submitted 2025-04-18; First posted 2025-04-25 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-04

CONDITIONS: Gastroesophageal Reflux Disease
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — flupentixol, melitracen drug combination; Lansoprazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients were treated with Flupentixol-Melitracen (FM) plus lansoprazole for 2 weeks (Experimental)
  Interventions: Drug: Flupentixol-Melitracen + Lansoprazole
- Patients were treated with placebo plus lansoprazole for 2 weeks (Placebo Comparator)
  Interventions: Drug: Lansoprazole and placebo

INTERVENTIONS:
Drug: Flupentixol-Melitracen + Lansoprazole — Flupentixol-Melitracen and Lansoprazole for the treatment of GERD
  Arms: Patients were treated with Flupentixol-Melitracen (FM) plus lansoprazole for 2 weeks
Drug: Lansoprazole and placebo — Placebo and Lansoprazole for GERD
  Arms: Patients were treated with placebo plus lansoprazole for 2 weeks

SUMMARY:
Gastroesophageal reflux disease (GERD) is a common chronic digestive system disorder with a high prevalence and a notably increasing trend. It imposes significant costs in terms of treatment expenses and impacts patients' quality of life. Acid suppression remains the primary treatment for GERD. However, numerous clinical studies have shown that 20-30% of patients still exhibit poor response to proton pump inhibitors (PPIs) even after completing a standard course of acid-suppressive therapy. Many studies have demonstrated that the incidence of abnormal psychological conditions, such as anxiety, depression, and obsessive-compulsive disorder, is higher in GERD patients compared to the general population. Current international consensus acknowledges that the application of psychosomatic medicine principles and the use of neuromodulators can effectively alleviate symptoms in patients with gut-brain interaction disorders. Nevertheless, with the growing emphasis on digestive-psychosomatic-holistic medicine in clinical practice and the deepening of research on "gut-brain interactions," recent studies in the field of psycho-gastroenterology have challenged the notion that psychological processes are unique to gut-brain interaction disorders. Instead, these processes may play a universal role in symptom generation across the entire spectrum of GERD. Previous experiments have confirmed that Flupentixol-Melitracen (FM) can improve symptoms in GERD patients with a low incidence of adverse reactions. Therefore, we aim to verify the efficacy and safety of neuromodulators in patients with GERD, reduce healthcare costs, and provide new insights for optimizing treatment strategies for GERD patients in the future.

ELIGIBILITY:
Inclusion Criteria:

- Adults aged 18-70 years with gastroesophageal reflux disease (GERD) meeting diagnostic criteria.

Exclusion Criteria:

* Patients with organic gastrointestinal disorders (e.g., celiac disease, inflammatory bowel disease, history of gastrointestinal malignancies);

Severe dysfunction of major organs (e.g., class IV cardiac dysfunction, hepatic failure, uremia, respiratory failure) or congenital diseases (e.g., hemophilia, Wilson's disease);

Hypersensitivity to study medications;

Patients who are pregnant, lactating, or planning pregnancy;

Use of monoamine oxidase inhibitors (e.g., linezolid or intravenous methylene blue) within the past 5 weeks;

Severe psychological symptoms or cognitive impairment (GAD-7 >15 or PHQ-9 ≥15);

Circulatory failure, central nervous system depression (e.g., acute alcohol, barbiturate, or opioid intoxication), or coma.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2025-04-24 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-10-30 (Actual)

PRIMARY OUTCOMES:
GERD questionnaire (GerdQ) | Until the end of the study, up to 12 weeks
  The GerdQ Scale is a validated tool for assessing gastroesophageal reflux disease (GERD). It includes 6 items evaluating symptom frequency (heartburn, regurgitation), extra-esophageal manifestations, and quality of life impact (e.g., sleep disturbance, medication use) over the past week. Scores range 0-18; ≥8 suggests high GERD likelihood, guiding stepwise treatment (lifestyle changes or PPIs).

CONTACTS AND LOCATIONS:
Overall Officials: Sheng L Chen, doctor, Principal Investigator — Shanghai Jiao Tong University School of Medicine，Renji Hospital
Locations (1):
- Shanghai Jiaotong university，renji hospital, Shanghai, Shanghai Municipality, China